CLINICAL TRIAL: NCT02422537
Title: The Effect of One Single Dose of Different Bran-based Dietary Platforms on the Colon Metabolism - A Study With (Stable) Isotopes in Healthy Volunteers
Brief Title: Effect of Different Bran-based Dietary Platforms on the Colon Metabolism in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ML11202
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Unmodified wheat bran (Active Comparator): One single dose om 20 g
  Interventions: Dietary Supplement: Unmodified wheat bran
- Wheat bran with reduced particle size (Active Comparator): One single dose of 20 g
  Interventions: Dietary Supplement: Wheat bran with reduced particle size
- Destarched pericarp-enriched wheat bran (Active Comparator): One single dose of 20 g
  Interventions: Dietary Supplement: Destarched pericarp-enriched wheat bran
- No bran-based dietary platform (Other): No wheat bran fractions is administered
  Interventions: Dietary Supplement: No wheat bran fraction

INTERVENTIONS:
Dietary Supplement: Unmodified wheat bran
  Arms: Unmodified wheat bran
Dietary Supplement: Wheat bran with reduced particle size
  Arms: Wheat bran with reduced particle size
Dietary Supplement: Destarched pericarp-enriched wheat bran
  Arms: Destarched pericarp-enriched wheat bran
Dietary Supplement: No wheat bran fraction
  Arms: No bran-based dietary platform

SUMMARY:
During this project the effect of 3 different bran-based dietary platforms on the fermentation on a readily fermentable substrate will be investigated using stable isotope techniques.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged between 18 and 65 years
* BMI between 18 and 27 kg/m²
* Stable eating pattern (3 meals/day on at least 5 days/week)

Exclusion Criteria:

* Use of antibiotics in the month preceding the study
* Abdominal surgery (except from appendectomy)
* Use of medication that affects the gastrointestinal tract during the last 2 weeks prior to the study including spasmolytics, anti-diarrhoea medication, anti-constipation medication
* Use of pre- or probiotic supplements in the month preceding the study
* Chronic gastrointestinal diseases, such as inflammatory bowel disease (Crohn's disease, ulcerative colitis), irritable bowel disease…
* Pregnancy or lactation
* Blood donation in the last 3 months
* Abnormal Hb-level (Standard range between 14 and 18 g/dL for men and between 12 and 16 g/dL for women)
* Participation in clinical studies involving radiation exposure in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quantification of acetate, propionate and butyrate production in the colon after consumption of each bran-based dietary platform | 2 years

SECONDARY OUTCOMES:
Estimation of the site of fermentation of a readily fermentable carbohydrate in the presence of different bran-based dietary platforms | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven/ UZ Leuven, Leuven, Vlaams-Brabant, Belgium